CLINICAL TRIAL: NCT00092222
Title: Targeted Oncolytic Virotherapy and Natural History Study of KSHV-Associated Multicentric Castleman's Disease With Laboratory and Clinical Correlates of Disease Activity
Brief Title: Virotherapy and Natural History Study of KHSV-Associated Multricentric Castleman s Disease With Correlates of Disease Activity
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 040275; 04-C-0275; NCT00099073 (obsolete NCT alias)
Record Dates: First submitted 2004-09-21; First posted 2004-09-22 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-27

CONDITIONS: Lymphoproliferative Disorder; HHV-8; Malignancy; HIV
Keywords: HHV-8; HIV; Malignancy; Lymphoproliferation; Lymph Node Hyperplasia; Multicentric Castleman DIsease; MCD; KSHV-MCD; KSHV Associated MCD; HIV Infections; Herpes Viruses
MeSH Terms: conditions — Lymphoproliferative Disorders; Neoplasms; Lymphadenopathy; Multi-centric Castleman's Disease; Macular dystrophy, corneal type 1; HIV Infections | interventions — Etoposide; Interferon-alpha; Rituximab; Zidovudine; liposomal doxorubicin; Bortezomib; Valganciclovir; Doxorubicin; Vincristine; Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; Prednisone; Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Active Treament 3 (Active Comparator): Patients not responding to high- dose zidovudine and valganciclovir alone may be treated with botezomib plus high- dose zidovudine and valganciclovir
  Interventions: Drug: Zidovudine; Drug: Bortezomib; Drug: Valganciclovir
- Active Treatment 1 (Active Comparator): Single agent sirolimus for patients where targeted oncolytic virotherapy seems suboptimal
  Interventions: Drug: Sirolimus
- Active Treatment 2 (Active Comparator): EPOCH chemotherapy with rituximab may be utilized to rescue such patients, with the intent of stabilizing suchpatients
  Interventions: Drug: Etoposide; Drug: Rituximab; Drug: Doxorubicin; Drug: Vincristine; Drug: Cyclophosphamide; Drug: Filgrastim (G-CSF); Drug: Prednisone
- Active Treatment 4 (Active Comparator): Rituximab with liposomal doxorubicin (R-Dox) followed by consolidation or lmaintenancel therapy with dose escalating interferon-alpha
  Interventions: Drug: Interferon-alpha; Drug: Rituximab; Drug: Liposomal Doxorubicin
- Active Treatment 5 (Active Comparator): High dose zidovudin and valganciclovir
  Interventions: Drug: Zidovudine; Drug: Valganciclovir
- Natural History (Active Comparator): Observation Only
  Interventions: Other: Observation Only

INTERVENTIONS:
Drug: Etoposide — Etoposide 50 mg/m2 /day continuous intravenous infusion (CIVI) over 24 hours x 4 days (days 1-4) of 21 day cycle. A maximum of 6 cycles of R-EPOCH-R will be administered except in exceptional circumstances.
  Arms: Active Treatment 2
Drug: Interferon-alpha — Ages 18 and over: Initial dose of 7.5 million units subcutaneous, three times weekly x 14 days; subsequent dosesincrease dose as tolerated each 14 days to a maximum of 45 million units subcutaneous three times weekly; Ages 12-17: Initial dose of 5 million units/m2 subcutaneous, three times weekly x 14 days Subsequent doses: Increase dose as tolerated each 14 days to a maximum of 30 million units/m2 subcutaneous, three times weekly
  Arms: Active Treatment 4
Drug: Rituximab — Rituximab 375 mg/m2 IV day 1, shall be administered prior to Doxil injection. When combined with EPOCH chemotherapy, Rituximab will be given on days 1 and 5.
  Arms: Active Treatment 2; Active Treatment 4
Drug: Zidovudine — Cycle 1: Zidovudine 600 mg PO QID x 7-21 days in outpatient setting;600 mg PO q6hours x 7-21 (Intravenous zidovudine 300 mg q 6 hours may be substituted) days for inpatients; Cycle 2 and beyond: 600 mg PO QID x 7 days in outpatient setting; 600 mg PO q 6 hours x 7 days (300 mg q 6 hours may be substituted)
  Arms: Active Treament 3; Active Treatment 5
Drug: Liposomal Doxorubicin — 21 day cycle; 20 mg/m2 Liposomal Doxorubicin given on day 1 and shall be administered after completion of Rituximab infusion from 2 to 6 cycles.
  Arms: Active Treatment 4
Drug: Bortezomib — 1.3 mg/m2 IV days 1, 4, 8, and 11. Cycle length is 21 days.
  Arms: Active Treament 3
Drug: Valganciclovir — Cycle 1: Valganciclovir 900 mg PO BID x 7-21 days in outpatient setting; 900 mg PO q 12 hours x 7-21 days for inpatients; Cycle 2 and beyond: 900 mg PO BID x 7 days for outpatients; 900 mg PO q 12 hours x 7 days (Intravenous ganciclovir 5 mg/kg may be substituted) for inpatients
  Arms: Active Treament 3; Active Treatment 5
Drug: Doxorubicin — 10 mg/m2 /day CIVI over 24 hours x 4 days (days 1-4) of 21 day cycle.
  Arms: Active Treatment 2
Drug: Vincristine — 0.4 mg/m2 /day CIVI over 24 hours x 4 days (days 1-4) of 21 day cycle.
  Arms: Active Treatment 2
Drug: Cyclophosphamide — Cyclophosphamide: if CD4 < 100 cells/mm3, 187 mg/m2 IV (Day 5) if CD4 greater than or equal to 100 cells/mm3, 375 mg/m2 IV (Day 5) of 21 day cycle.
  Arms: Active Treatment 2
Drug: Filgrastim (G-CSF) — Filgrastim 300 micrograms subcutaneous daily beginning day 6 until absolute neutrophil count recovery 5000 cells/mm3 (Pegfilgrastim may be substituted with PI approval, at the recommended dose of one 6mg syringe)
  Arms: Active Treatment 2
Drug: Prednisone — Prednisone 60 mg/m2/day PO x 5 days (days 1-5)of 21 day cycle.
  Arms: Active Treatment 2
Drug: Sirolimus — Maximum daily dose of 40 mg given as a single agent on 21 day cycle.
  Arms: Active Treatment 1
Other: Observation Only — Observation of symptoms
  Arms: Natural History

SUMMARY:
This study will gain information about a rare disorder called KSHV-associated multicentric Castleman's disease (MCD). KSHV, a virus, causes several kinds of cancer, including some forms of MCD. KSHV stands for the Kaposi's sarcoma herpes virus, also called human herpes virus-8, or HHV-8. Researchers want to understand the biology of KSHV-MCD to identify how this disease causes illness and to find ways to treat it. There is no standard therapy effective for all cases of KSHV-MCD. The disease is often fatal, and about half the people who have it die within 2 years of diagnosis.

Participants ages 18 and older may be eligible for this study. Participation entails more drawing of blood and having repeated tumor biopsies than if patients received treatment in a non-research setting. Researchers would like to learn more about the relationship of KSHV and Castleman's disease symptoms, and they want to obtain at least three biopsies in this study.

There are some side effects of experimental therapy that participants may take for KSHV-MCD. Zidovudine, or Retrovir(R), is used at a high dose. It is given orally or through a vein, four times daily, for 7 days or longer. Zidovudine can cause nausea, vomiting, decreased bone marrow function, and decreased blood counts. Combined with valganciclovir, or Valcyte(TM), it is likely to be more toxic to bone marrow. Valganciclovir can cause problems with bone marrow function, leading to low blood counts, sterility, and defects in a fetus. Combined with zidovudine, valganciclovir may cause more toxicity to the bone marrow. It is given twice daily for 7 days or longer. Bortezomib, or Velcade(TM), is given for a few seconds by a rapid push through a needle into the vein. It is given twice weekly for four doses and then stopped for 1 week. Bortezomib can sometimes cause low blood pressure; it also can cause gastrointestinal problems and a low blood platelet count. Rituximab and liposomal doxorubicin are drugs given by a catheter into a vein. Interferon-alpha is given by injection into the skin. Those drugs are not experimental, but their use in Castleman's disease is experimental.

Some participants may be treated with a combination of chemotherapy followed by interferon-alpha. Interferon-alpha is infected into the skin by a needle. The natural form of interferon is produced by the body and helps to control viral infections. KSHV decreases the effect of the body's interferon, and the researchers want to see if giving higher doses of interferon will help to control KSHV infection.

A positron emission tomography (PET) scan, for research purposes only, may be done up to three times a year. A radioactive sugar molecule called fluorodeoxyglucose, or FDG, is used. It is believed that activated lymphocytes that may be found in participants' disease might use more FDG because these cells burn more glucose fuel.

This study may or may not have a direct benefit for participants. However, detailed assessments made throughout the study may provide information to help the doctors treat KSHV-MCD better.

DETAILED DESCRIPTION:
Background:

* Multicentric Castleman's disease (MCD) is a rare but lethal Kaposi's sarcoma-associated herpesvirus (KSHV) associated lymphoproliferative disorder with a median survival of 2 years. It occurs more often in HIV-infected individuals than those without HIV infection. The poor prognosis is not fully explained by the underlying HIV, as the HIV-negative cases appear to have no survival advantage over the HIV-positive cohort. The disease has no defined standard treatment and has not been prospectively studied in a comprehensive manner.
* KSHV-MCD may provide a model for the development of targeted oncolytic virotherapy or other pathogenesis-based approaches to viral-associated malignancies. In KSHV-MCD, viral encoded kinase genes appear to be possible targets to exploit in a virotherapy approach. Specific viral encoded genes appear to convert zidovudine and ganciclovir (or valganciclovir) into toxic phosphorylated moieties within the KSHV-infected tumor cells, to specifically target the KSHV-infected cells thus leading to specific cell death. If successful, this could have direct therapeutic benefit to participants and also provide a model for further development of this approach in other tumors.

Objectives

-To study and describe the natural history of KSHV-MCD.

Eligibility

* Age >= 18 years
* Biopsy proven KSHV-associated MCD

Design

* Natural History study
* Inclusion of treatment as needed, with guidelines for preliminary investigation of a variety of specific treatments of interest

  * High-dose zidovudine and ganciclovir
  * High-dose zidovudine and ganciclovir and bortezomib
  * Sirolimus
  * Rituximab with liposomal doxorubicin followed by interferon-alpha or high-dose AZT with valganciclovir
  * Rituximab with EPOCH chemotherapy

ELIGIBILITY:
* INCLUSION CRITERIA:

Age greater than or equal to 18 years.

Biopsy proven KSHV-associated MCD, confirmed in the Laboratory of Pathology, CCR.

Willing to give informed consent.

EXCLUSION CRITERIA:

Any abnormality that would be scored as NCI CTCAE v 3.0 Grade IV toxicity that is unrelated to HIV, its treatment, or to MCD that would preclude protocol treatment and/or observation only.

Presence of another malignancy requiring current treatment that would preclude the use of all of the study treatments or the ability to monitor the natural history of MCD untreated.

Pregnant women are excluded from this study as certain of the study agents have the potential for teratogenic effects

Any condition or set of circumstances that in the opinion of the investigators would make participation in this study unsafe or otherwise inappropriate for a given individual.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-10-28 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Describe natural history | Study Closure
  Response to treatment

SECONDARY OUTCOMES:
overall survival | Study Closure
  percentage of patients alive until study closure
Number of flares | Study closure
  Quantify the number of flares requiring treatment in patients enrolled in this study

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Oksenhendler E, Carcelain G, Aoki Y, Boulanger E, Maillard A, Clauvel JP, Agbalika F. High levels of human herpesvirus 8 viral load, human interleukin-6, interleukin-10, and C reactive protein correlate with exacerbation of multicentric castleman disease in HIV-infected patients. Blood. 2000 Sep 15;96(6):2069-73. PMID 10979949
- [Background] Gaidano G, Capello D, Pastore C, Antinori A, Gloghini A, Carbone A, Larocca LM, Saglio G. Analysis of human herpesvirus type 8 infection in AIDS-related and AIDS-unrelated primary central nervous system lymphoma. J Infect Dis. 1997 May;175(5):1193-7. doi: 10.1086/593456. PMID 9129084
- [Background] Oksenhendler E, Duarte M, Soulier J, Cacoub P, Welker Y, Cadranel J, Cazals-Hatem D, Autran B, Clauvel JP, Raphael M. Multicentric Castleman's disease in HIV infection: a clinical and pathological study of 20 patients. AIDS. 1996 Jan;10(1):61-7. PMID 8924253
- [Derived] Lage SL, Ramaswami R, Rocco JM, Rupert A, Davis DA, Lurain K, Manion M, Whitby D, Yarchoan R, Sereti I. Inflammasome activation in patients with Kaposi sarcoma herpesvirus-associated diseases. Blood. 2024 Oct 3;144(14):1496-1507. doi: 10.1182/blood.2024024144. PMID 38941593
- [Derived] Ramaswami R, Lurain K, Polizzotto MN, Ekwede I, Waldon K, Steinberg SM, Mangusan R, Widell A, Rupert A, George J, Goncalves PH, Marshall VA, Whitby D, Wang HW, Pittaluga S, Jaffe ES, Little RF, Uldrick TS, Yarchoan R. Characteristics and outcomes of KSHV-associated multicentric Castleman disease with or without other KSHV diseases. Blood Adv. 2021 Mar 23;5(6):1660-1670. doi: 10.1182/bloodadvances.2020004058. PMID 33720337
- [Derived] Uldrick TS, Polizzotto MN, Aleman K, Wyvill KM, Marshall V, Whitby D, Wang V, Pittaluga S, O'Mahony D, Steinberg SM, Little RF, Yarchoan R. Rituximab plus liposomal doxorubicin in HIV-infected patients with KSHV-associated multicentric Castleman disease. Blood. 2014 Dec 4;124(24):3544-52. doi: 10.1182/blood-2014-07-586800. Epub 2014 Oct 20. PMID 25331113
- [Derived] Polizzotto MN, Uldrick TS, Wang V, Aleman K, Wyvill KM, Marshall V, Pittaluga S, O'Mahony D, Whitby D, Tosato G, Steinberg SM, Little RF, Yarchoan R. Human and viral interleukin-6 and other cytokines in Kaposi sarcoma herpesvirus-associated multicentric Castleman disease. Blood. 2013 Dec 19;122(26):4189-98. doi: 10.1182/blood-2013-08-519959. Epub 2013 Oct 30. PMID 24174627
- [Derived] Uldrick TS, Polizzotto MN, Aleman K, O'Mahony D, Wyvill KM, Wang V, Marshall V, Pittaluga S, Steinberg SM, Tosato G, Whitby D, Little RF, Yarchoan R. High-dose zidovudine plus valganciclovir for Kaposi sarcoma herpesvirus-associated multicentric Castleman disease: a pilot study of virus-activated cytotoxic therapy. Blood. 2011 Jun 30;117(26):6977-86. doi: 10.1182/blood-2010-11-317610. Epub 2011 Apr 12. PMID 21487108
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0275.html